CLINICAL TRIAL: NCT04240626
Title: Multimodal Analgesia Effect on Post Surgical Patient
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1452523
Record Dates: First submitted 2019-10-16; First posted 2020-01-27 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Obesity, Morbid; Surgery; Bariatric Surgery Candidate
Keywords: Bariatric Surgery,; Pain Control; Gabapentinin
MeSH Terms: conditions — Obesity, Morbid; Agnosia | interventions — Gabapentin; Hydromorphone; Oxycodone; oxycodone-acetaminophen; Hydrocodone; Ondansetron; Scopolamine; Lorazepam; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Patients will receive Gabapentin and Ofirmev post surgery (dosage based on patients pre-operative weight) with on-call medications as needed including narcotic analgesia for breakthrough pain control
Masking Description: Patients agreeing to participate in the study will be assigned one of two treatment arms. Neither the care team nor the patient will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): The group will receive the standard of care pain control protocol after index Bariatric Surgery which includes the use of a PCA (patient controlled analgesia) with Dilaudid or Morphine Sulphate, transitioning to oral narcotic based pain control medications.
  Interventions: Drug: Dilaudid Injectable Product; Drug: Marcaine Injectable Product; Drug: Oxycodone Hydrochloride; Drug: Hycet 7.5Mg-325Mg/15Ml Solution; Drug: Zofran Injection; Drug: Scopolamine patch; Drug: Ativan; Drug: Flexeril Oral Product
- Multi-Modal (Experimental): Patients will receive Gabapentin pre-operatively on-call 120 minutes prior to surgery starting. Patients at the conclusion of surgery will have additional doses of Ofirmev (IV Tylenol) and Gabapentin via IV based on patients pre-operative weight. Post surgery the patient will be transitioned to oral pain medications (Tylenol and Gabapentin) with rescue medications available for breakthrough pain control.
  Interventions: Drug: Neurontin; Drug: Dilaudid Injectable Product; Drug: Marcaine Injectable Product; Drug: Oxycodone Hydrochloride; Drug: Hycet 7.5Mg-325Mg/15Ml Solution; Drug: Zofran Injection; Drug: Scopolamine patch; Drug: Ativan; Drug: Flexeril Oral Product; Drug: Tylenol Suspension

INTERVENTIONS:
Drug: Neurontin — 600 mg on-call prior to surgery, post surgery 100 mg liquid q 8-12 hours post surgery with Tylenol every 6 hours
  Other Names: Gabapentin
  Arms: Multi-Modal
Drug: Dilaudid Injectable Product — .5-1 mg IV Q3 hours and IV Tylenol 1000mg every 6 hours post surgery transitioning to oral pain control medications (Hycet 7.5/325mg/5 ml, 5-10 ml every 4 hours
  Other Names: Hydromorphone
Drug: Marcaine Injectable Product — 0.25% local injectable anesthetic agent infiltrated at all laparoscopic incision sites for both groups.
Drug: Oxycodone Hydrochloride — 1 mg/ml oral solution, dosage 5-10mg q4h prn for pain control
Drug: Hycet 7.5Mg-325Mg/15Ml Solution — Dosage: 10-15ml q4h prn for pain control
  Other Names: Hydrocodone
Drug: Zofran Injection — 4 mg IV for nausea control while inpatient, prn
  Other Names: Odanesetron
Drug: Scopolamine patch — Topical application patch for nausea control, used with/without Ativan.
  Other Names: Scopolamine
Drug: Ativan — 0.5mg IV as needed in conjunction with/without Scopolamine and Zofran for Nausea control
Drug: Flexeril Oral Product — 5 mg orally q8h prn for muscle spasms.
  Other Names: Cyclobenziparin
Drug: Tylenol Suspension — 1000 mg q6h PRN for pain control.
  Other Names: Acetaminophen
  Arms: Multi-Modal

SUMMARY:
Patients undergoing Bariatric Surgery at the University of California Davis Medical Center will be divided into two groups, one receiving Standard of Care pain control medications vs the second group which will receive non-narcotic pain medications with rescue pain medications available if needed

DETAILED DESCRIPTION:
Pain control after weight loss surgery is challenging due to the alteration of digestive system anatomy and limitation on using medications which can either be crushed or in liquid form for the first 10 days to 14 days after surgery. Additionally there are multiple programs in place to eliminate the use of narcotic/opioid based pain medications due their potential addictive risks.

This study compares two groups of patients whom will have Roux en Y Gastric Bypass Surgery at UC Davis Medical Center, the control group will receive standard of care pain control medications (including opioid based medications) compared to the research arm, this group will receive Gabapentinin and Tylenol for pain control after surgery with rescue pain medications available if needed.

Post surgery both groups will be managed by the Bariatric Surgery Team and will be contacted periodically as part of the standard of care to monitor pain control and usage of any rescue medications (if needed).

ELIGIBILITY:
Inclusion Criteria:

* Women who undergo index weight loss procedures at UC Davis Medical Center
* Women with a BMI =>30
* Age from 35-65
* American Society of Anesthesiology (ASA) score of 3 or less
* No previous history of prior abdominal/foregut surgery

Exclusion Criteria:

* Not having an index weight los surgery for obesity
* Do not meet the NIH Standards for weight loss surgery
* Additional planned or unplanned procedures during the index surgical procedure such as Cholecystectomy or extensive lysis of adhesions (>30 minutes)
* BMI < 30
* Men
* Women considering or currently planning on gender altering/modification
* ASA score of 4 or higher
* Patients less than 35 years of age or older than 65 years of age at the time of surgical consent
* A history of open abdominal surgery including umbilical, ventral, or splengalic hernia repair with or without mesh implantation, transplant or vascular surgery or any foregut procedures including hiatal hernia repair or anti-reflux surgery
* Arthritis, Fibromyalgia, chronic pain syndrome
* Other conditions requiring daily use of oral pain medications
* Prisoners
* Allergy to Gabapentin

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
Change In Post Operative Pain Intensity | 3 Days and 14 Days Post Surgery
  Using the Wong-Baker Pain Rating Scale-0=No Pain, 2-4, Slight Pain, 6-8, Moderate Pain, 9-10, Severe Pain
Change in Oral Morphine Equivalence (OME) from 3 days and 14 days post surgery | 3 Days and 14 Days Post Surgery
  OME Table is used to measure opioid use post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R Ali, MD, FACS, Principal Investigator — Professor of Surgery; Barbara Jachniewicz, MSN, CRNFA,, Principal Investigator — Nurse Practitioner, Department of Surgery
Locations (1):
- UC Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No